CLINICAL TRIAL: NCT06972576
Title: Clinical Study of Combined EphA2-targeted CAR-DC and CAR-T Cell Therapy for Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0164
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Chimeric Antigen Receptor Dendritic Cells; Chimeric Antigen Receptor T-Cells; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T and CAR-DC Combination Therapy (Experimental): This arm involves the sequential administration of two biological interventions with EphA2-targeted CAR-DCs administered first, followed by EphA2-targeted CAR-T cells.
  Interventions: Biological: EphA2-targeted CAR-T Cells; Biological: EphA2-targeted CAR-DCs

INTERVENTIONS:
Biological: EphA2-targeted CAR-T Cells — Autologous T cells genetically modified to express a chimeric antigen receptor (CAR) targeting EphA2
Biological: EphA2-targeted CAR-DCs — Autologous dendritic cells (DCs) genetically modified to express a chimeric antigen receptor (CAR) targeting EphA2

SUMMARY:
This is an open-label, single-arm clinical study designed to evaluate the safety and preliminary efficacy of EphA2-targeted CAR-DC combined with CAR-T cell therapy in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Main purpose:

To evaluate the safety of EphA2-targeted CAR-T cells in combination with CAR-DCs in patients with advanced non-small cell lung cancer during the dose-escalation phase.

To determine the maximum tolerated dose of EphA2-targeted CAR-DCs when administered in combination with CAR-T cells.

Secondary purpose:

To assess the overall response rate (ORR), including complete response (CR) and partial response (PR), as well as overall survival (OS) and disease-free survival (DFS) in patients receiving the combination therapy.

To evaluate the in vivo persistence, immunophenotype, and functional activity of CAR-T cells and CAR-DCs following infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed stage IV non-small cell lung cancer (NSCLC) with at least one measurable lesion according to RECIST 1.1 criteria (i.e., a lesion with the longest diameter ≥10 mm on spiral CT scan or a lymph node with a short axis ≥15 mm).
2. Tumor tissue tested positive for EphA2 expression by immunohistochemistry (≥20%).
3. Disease progression after standard treatment or no available standard treatment (patients must have received at least two prior systemic therapies, including but not limited to chemotherapy and immune checkpoint inhibitors; patients with actionable driver mutations must have failed targeted therapy).
4. ECOG performance status: 0-1.
5. Expected survival ≥6 months.
6. Toxicities related to prior anti-tumor treatments must have resolved to baseline levels or ≤ Grade 1 (excluding residual alopecia); Grade ≤2 neurotoxicity is acceptable. Washout periods: 4 weeks for chemotherapy and immunotherapy, 2 weeks for targeted therapy.
7. Adequate organ function, including:

   * Adequate hematologic function: Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥75×10^9/L, hemoglobin ≥9 g/dL. No transfusions, granulocyte colony-stimulating factor (G-CSF), thrombopoietin, or erythropoietin allowed within 14 days before blood tests.
   * Adequate hepatic function: Total bilirubin (TBIL) <1.5× upper limit of normal (ULN); AST and ALT <2.5×ULN. For patients with Gilbert's syndrome, TBIL <2×ULN; if liver metastases are present, AST and ALT <5×ULN.
   * Adequate renal function: Serum creatinine (Cr) ≤1.5×ULN, or if Cr >1.5×ULN, creatinine clearance (CrCl) ≥60 mL/min calculated using the Cockcroft-Gault formula.
   * Adequate coagulation function: Prothrombin time (PT) and activated partial thromboplastin time (APTT) <1.5×ULN; international normalized ratio (INR) <1.5 or within the target range if on anticoagulant therapy.
8. Subjects of reproductive potential must be willing to use effective contraception.
9. Ability to understand and voluntarily sign the informed consent form.
10. Willingness to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Pathologically confirmed mixed histology, such as adenosquamous carcinoma of the lung.
2. Tumor-related emergencies requiring urgent treatment, such as malignant pericardial effusion or cardiac tamponade, superior vena cava syndrome, or spinal cord compression.
3. Significant cardiovascular diseases, including:

   * Documented cardiovascular events within the past 6 months, such as myocardial infarction, angina, heart failure, severe arrhythmia, or having undergone angioplasty, stent implantation, or coronary artery bypass surgery.
   * Clinically significant QT/QTcF prolongation (QT/QTcF > 470 ms in females or > 450 ms in males).
4. Clinically significant bleeding tendency or coagulation disorders, such as hemophilia.
5. HIV or syphilis infection; active hepatitis B or C:

   * Hepatitis B: HBV-DNA ≥ 1000 IU/mL.
   * Hepatitis C: Positive HCV RNA with abnormal liver function.
6. History of involuntary commitment due to psychiatric disorders or other psychological conditions deemed unsuitable for treatment by the investigator.
7. Presence of other autoimmune diseases, or long-term use of immunosuppressive agents or corticosteroids.
8. Poor medication compliance.
9. Any other condition that the investigator considers grounds for exclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 3 month post CAR-T cells and CAR-DCs infusion
  To evaluate adverse events occurring within the first three months following infusion of EphA2-targeted CAR- T cells and CAR-DCs. The assessment includes incidence and severity of treatment-related symptoms such as neurological toxicity, hematological abnormalities, infections, autoimmune reactions, and secondary malignancies.
Efficacy: Remission Rate | 3 months post CAR-T cells and CAR-DCs infusion
  To evaluate the proportion of participants who achieve an objective tumor response, including complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
Progression-Free Survival | Up to 24 months post CAR-T cells and CAR-DCs infusion
Overall Survival | Up to 24 months post CAR-T cells and CAR-DCs infusion
Relapse Rate | Up to 24 months post CAR-T cells and CAR-DCs infusion
Duration of Response | Up to 24 months post CAR-T cells and CAR-DCs infusion
In Vivo Persistence of CAR-T cells and CAR-DCs and Cytokine Profile Monitoring | First 2 weeks post CAR-T cells and CAR-DCs infusion
  The copy number of CAR-T cells and CAR-DCs in PBMCs will be measured by qPCR to assess in vivo persistence.
  Serum cytokine levels, including IL-2, IL-4, IL-6, IFN-γ, TNF-α, IL-10, IL-12, and IL-17A, will be quantified by ELISA to evaluate immune activation following cell infusion.
Objective Response Rate in Participants Receiving Different Doses of CAR-DCs | Up to 24 months post CAR-T cells and CAR-DCs infusion
  The proportion of participants in each CAR-DCs dose cohort (5x10^6, 1x10^7, 3x10^7, and 9x10^7 cells) who achieve an objective tumor response, including completeremission (CR) or partial remission (PR). All participants received a fixed dose of EphA2-targeted CAR-T cells (2x10^6 cells/kg) following CAR-DCs infusion.
Incidence and Severity of Treatment-Related Adverse Events in Participants Receiving Different Doses of CAR-DCs | Up to 24 months post CAR-T cells and CAR-DCs infusion
  To evaluate adverse events occurring following infusion of EphA2-targeted CAR-DCs and CAR-T cells. Participants will receive CAR-DCs at one of four dose levels (5x10^6, 1x1 0^7, 3x10^7, and 9x10^7 cells), followed by a fixed dose of EphA2-targeted CAR-T cells(2x10^6 cells/kg). The assessment includes the incidence and severity of treatment-related symptoms such as neurological toxicity, hematological abnormalities, infections, autoimmune reactions, and secondary malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China